CLINICAL TRIAL: NCT03890510
Title: Effect of Different Fluid Volume on Ocular Parameters in Patients Undergoing Spine Surgery in Prone Position
Brief Title: The Effect of High vs. Low Fluid Volume on Ocular Parameters in Prone Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Yu Yang, MD, Principal Investigator, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FOCUS
Record Dates: First submitted 2019-02-21; First posted 2019-03-26 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Prone Position; Blood Volume; Intraocular Pressure
Keywords: pulse pressure variation; intraocular pressure; optic sheath diameter; spine surgery; prone position
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to the limited fluid infusion group and the loose fluid infusion group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low PPV Group (Active Comparator): After anesthesia induction, patients will receive spine surgery under general anesthesia in the prone position. Ringer's lactate solution will be infused at 1ml/（kg·h ） as a basal speed. Ringer's lactate solution at a volume of 250ml will be used as a bolus dose. Repeat bolus doses will be given to maintain PPV at 6~9% when necessary. Intraoptic pressure and optic sheath diameter will be measured at multiple time points.
  Interventions: Other: Ringer's Lactate solution; Procedure: Spine surgery under general Anesthesia in the prone position
- High PPV Group (Active Comparator): After anesthesia induction, patients will receive spine surgery under general anesthesia in the prone position. Ringer's lactate solution will be infused at 1ml/（kg·h ） as a basal speed. Ringer's lactate solution at a volume of 250ml will be used as a bolus dose. Repeat bolus doses will be given to maintain PPV at 13~16% when necessary. Intraoptic pressure and optic sheath diameter will be measured at multiple time points.
  Interventions: Other: Ringer's Lactate solution; Procedure: Spine surgery under general Anesthesia in the prone position

INTERVENTIONS:
Other: Ringer's Lactate solution — Patients in both groups will receive Ringer's lactate solution continuously during operation with different infusion volume.
Procedure: Spine surgery under general Anesthesia in the prone position — The surgery, general anesthesia, and the placement of the prone position will be performed according to the standard procedures.

SUMMARY:
The purpose of this trial is to compare the effect of different fluid volume infusion on ocular parameters in patients undergoing spine surgery in prone position.

DETAILED DESCRIPTION:
In the prone position, the intraocular pressure and optic nerve sheath diameter increase progressively with time as compared with those in the supine position. Excessive fluid infusion may further increase intraocular pressure and optic nerve sheath diameter. Pulse pressure variation (PPV) is a dynamic index which can effectively assess fluid responsiveness during general anesthesia.Therefore,the investigators have designed a study to compare the effect of different fluid volume infusion guided by low and high PPV indices on intraocular pressure and optic nerve sheath of patients undergoing prone spine surgery with general anesthesia. One group of the patients will receive relatively loose fluid infusion (target value of PPV: 6%-9%),while the other group of the patients will receive limited fluid infusion (target value of PPV: 13%-16%).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective spine surgery in prone position under general anesthesia
* American Society of Anesthesiologists (ASA) physical status I or II
* Have signed consent form

Exclusion Criteria:

* History of eye disease or eye surgery
* Pregnancy or breast feeding
* Known Allergy to latex or Ringer's lactate solution
* Hyperlactacidemia，uncontrolled hypertension, diabetes mellitus, arrhythmia, cardiovascular disease，chronic pulmonary disease, swelling of any body part, abnormal of liver or renal function, anemia, etc.
* Body mass index（BMI）>30
* Expected operation time >6 hours
* Estimated Intraoperative hemorrhage >1000ml
* Taking part in other clinical trials in the last 3 months or at present

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
The change of intraocular pressure | 10min after anesthesia induction（supine1）, 10min after prone position(prone1), 1 hour after the prone position(prone2), 2 hour after the prone position(prone3),at the end of the surgery(prone4), and 10min after return to the supine position(supine2).
  Intraocular pressure will be measured with a TONO-PEN AVIA handheld tonometer.

SECONDARY OUTCOMES:
The change of the optic sheath diameter | 10min after anesthesia induction（supine1）, 10min after prone position(prone1), 1 hour after the prone position(prone2), 2 hour after the prone position(prone3),at the end of the surgery(prone4), and 10min after return to the supine position(supine2).
  The optic sheath diameter will be measured with a Sonocite Portable Ultrasonic System EDGE.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Yang, M.D., Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng MA, Todorov A, Tempelhoff R, McHugh T, Crowder CM, Lauryssen C. The effect of prone positioning on intraocular pressure in anesthetized patients. Anesthesiology. 2001 Dec;95(6):1351-5. doi: 10.1097/00000542-200112000-00012. PMID 11748391
- [Background] Uribe AA, Baig MN, Puente EG, Viloria A, Mendel E, Bergese SD. Current intraoperative devices to reduce visual loss after spine surgery. Neurosurg Focus. 2012 Aug;33(2):E14. doi: 10.3171/2009.8.FOCUS09151. PMID 22853832
- [Background] American Society of Anesthesiologists Task Force on Perioperative Visual Loss. Practice advisory for perioperative visual loss associated with spine surgery: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Visual Loss. Anesthesiology. 2012 Feb;116(2):274-85. doi: 10.1097/ALN.0b013e31823c104d. No abstract available. PMID 22227790
- [Background] Blecha S, Harth M, Schlachetzki F, Zeman F, Blecha C, Flora P, Burger M, Denzinger S, Graf BM, Helbig H, Pawlik MT. Changes in intraocular pressure and optic nerve sheath diameter in patients undergoing robotic-assisted laparoscopic prostatectomy in steep 45 degrees Trendelenburg position. BMC Anesthesiol. 2017 Mar 11;17(1):40. doi: 10.1186/s12871-017-0333-3. PMID 28284189
- [Background] Warner MA. Postoperative visual loss: experts, data, and practice. Anesthesiology. 2006 Oct;105(4):641-2. doi: 10.1097/00000542-200610000-00002. No abstract available. PMID 17006056
- [Background] Grant GP, Szirth BC, Bennett HL, Huang SS, Thaker RS, Heary RF, Turbin RE. Effects of prone and reverse trendelenburg positioning on ocular parameters. Anesthesiology. 2010 Jan;112(1):57-65. doi: 10.1097/ALN.0b013e3181c294e1. PMID 19996956
- [Background] Lee LA, Roth S, Posner KL, Cheney FW, Caplan RA, Newman NJ, Domino KB. The American Society of Anesthesiologists Postoperative Visual Loss Registry: analysis of 93 spine surgery cases with postoperative visual loss. Anesthesiology. 2006 Oct;105(4):652-9; quiz 867-8. doi: 10.1097/00000542-200610000-00007. PMID 17006060
- [Background] Lee LA. Perioperative visual loss and anesthetic management. Curr Opin Anaesthesiol. 2013 Jun;26(3):375-81. doi: 10.1097/ACO.0b013e328360dcd9. PMID 23614957
- [Background] Li A, Swinney C, Veeravagu A, Bhatti I, Ratliff J. Postoperative Visual Loss Following Lumbar Spine Surgery: A Review of Risk Factors by Diagnosis. World Neurosurg. 2015 Dec;84(6):2010-21. doi: 10.1016/j.wneu.2015.08.030. Epub 2015 Sep 1. PMID 26341434
- [Background] Nandyala SV, Marquez-Lara A, Fineberg SJ, Singh R, Singh K. Incidence and risk factors for perioperative visual loss after spinal fusion. Spine J. 2014 Sep 1;14(9):1866-72. doi: 10.1016/j.spinee.2013.10.026. Epub 2013 Nov 8. PMID 24216394
- [Background] Roth S. Perioperative visual loss: what do we know, what can we do? Br J Anaesth. 2009 Dec;103 Suppl 1(Suppl 1):i31-40. doi: 10.1093/bja/aep295. PMID 20007988
- [Result] Farag E, Sessler DI, Kovaci B, Wang L, Mascha EJ, Bell G, Kalfas I, Rockwood E, Kurz A. Effects of crystalloid versus colloid and the alpha-2 agonist brimonidine versus placebo on intraocular pressure during prone spine surgery: a factorial randomized trial. Anesthesiology. 2012 Apr;116(4):807-15. doi: 10.1097/ALN.0b013e3182475c10. PMID 22322966
- [Derived] Yang XY, Wei MM, Tan H, Wang HL, Luo MQ, Xu M, Wang YW. The effect of restrictive vs. liberal fluid protocols on ocular parameters in patients undergoing prone spine surgery: a randomized controlled trial. Perioper Med (Lond). 2023 Jun 12;12(1):23. doi: 10.1186/s13741-023-00310-6. PMID 37308905